CLINICAL TRIAL: NCT00983177
Title: Colchicine Treatment for Chronic Shoulder Pain Related to Calcific Tendonitis: Double Blind Placebo-controlled Study
Brief Title: Colchicine Treatment for Chronic Shoulder Pain Related to Calcific Tendonitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Gleb Slobodin, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: colchicine1
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Calcific Tendonitis
MeSH Terms: interventions — Colchicine; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- colchicine (Active Comparator)
  Interventions: Drug: Colchicine
- Lactose capsule (Placebo Comparator)
  Interventions: Drug: lactose

INTERVENTIONS:
Drug: Colchicine — 0.5 mg twice daily for 4 months
  Arms: colchicine
Drug: lactose — lactose capsules twice daily
  Arms: Lactose capsule

SUMMARY:
Chronic pain due to calcific tendonitis of shoulder is a prevalent condition usually treated with recurrent courses of NSAIDs, physical therapy or surgical interventions. Colchicine has been reported to be effective in the acute attack of shoulder tendonitis, however, has never been examined in controlled study in patients with chronic shoulder pain secondary to calcific tendonitis. Eighty patients with chronic shoulder pain (at least 3 months duration) due to calcific tendonitis will be randomized to receive colchicine 0.5 mg twice daily or placebo (lactose capsules) for 4 months. At the end of this blinded part of the study, patients who received placebo and did not improve, will be eligible to continue study in the open mode for additional 4 months with study drug. Efficacy (VAS for shoulder pain, shoulder range of motion and shoulder pain and disability index) and safety (blood tests) follow-ups will be scheduled bi-monthly for all patients.

ELIGIBILITY:
Inclusion Criteria:

* chronic, more than 3 months duration, shoulder pain
* tendinous calcifications on shoulder X-rays

Exclusion Criteria:

* renal insufficiency
* liver insufficiency
* lactose intolerance
* hypersensitivity to colchicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
VAS for shoulder pain | 4-8 months
shoulder range of motion | 4-8 months
shoulder pain and disability index | 4-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Rosner, MD, Study Director — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel